CLINICAL TRIAL: NCT04908488
Title: Clinical Performance of Two Daily Disposable Toric Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLA306-P001
Record Dates: First submitted 2021-05-28; First posted 2021-06-01 (Actual); Results first posted 2022-09-23 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: Refractive Errors; Ametropia; Astigmatism
Keywords: Contact Lenses; Disposable
MeSH Terms: conditions — Refractive Errors; Astigmatism

STUDY DESIGN:
Intervention Model Description: Subjects will receive treatment based upon the randomized treatment sequence assignment.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- P1fA, then AMfA (Other): Verofilcon A toric contact lenses worn first, with etafilcon A toric contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A toric contact lenses; Device: Etafilcon A toric contact lenses
- AMfA, then P1fA (Other): Etafilcon A toric contact lenses worn first, with verofilcon A toric contact lenses worn second, as randomized. Each study lens type will be worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
  Interventions: Device: Verofilcon A toric contact lenses; Device: Etafilcon A toric contact lenses

INTERVENTIONS:
Device: Verofilcon A toric contact lenses — Soft contact lenses for optical correction of astigmatism
  Other Names: PRECISION1™ for Astigmatism; P1fA
Device: Etafilcon A toric contact lenses — Soft contact lenses for optical correction of astigmatism
  Other Names: 1-DAY ACUVUE MOIST® for ASTIGMATISM; AMfA

SUMMARY:
The purpose of this study is to compare the clinical performance of PRECISION1™ for Astigmatism (P1fA) contact lenses with 1-DAY ACUVUE MOIST® for ASTIGMATISM (AMfA) contact lenses.

DETAILED DESCRIPTION:
Subjects will be expected to attend 4 visits and wear study lenses daily for at least 10 hours per day. The total duration of subject participation will be up to 22 days.

ELIGIBILITY:
Inclusion Criteria:

* Successful wear of toric soft contact lenses in both eyes for a a minimum of 5 days per week and 10 hours per day during the past 3 months.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Habitual PRECISION1 for Astigmatism or 1-DAY ACUVUE MOIST for ASTIGMATISM contact lens wearers.
* Any spherical monovision and multifocal lens wearers.
* Routinely sleeping in contact lenses for at least 1 night per week over the last 3 months prior to enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-22 (Actual); Study Completion 2021-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (8):
- United States (8):
  - Alcon Investigator 8135, Los Angeles, California
  - Alcon Investigator 8062, Oakland, California
  - Alcon Investigator 6355, Orlando, Florida
  - Alcon Investigator 6614, Franklin Park, Illinois
  - Alcon Investigator 6645, Shawnee Mission, Kansas
  - Alcon Investigator 3382, Wyomissing, Pennsylvania
  - Alcon Investigator 6353, Memphis, Tennessee
  - Alcon Investigator 2786, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 8 investigative sites located in the United States.
Pre-assignment Details: Of the 115 enrolled, 1 participant was exited from the study prior to randomization as a screen failure. This reporting group includes all subjects/eyes exposed to any study lenses evaluated in this study (114).
Units Other Than Participants: eyes
Groups:
- P1fA, Then AMfA: Verofilcon A toric contact lenses worn first, with etafilcon A toric contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
- AMfA, Then P1fA: Etafilcon A toric contact lenses worn first, with verofilcon A toric contact lenses worn second, as randomized. Each study lens type was worn bilaterally (in both eyes) for 8 -0/+3 days in a daily disposable modality.
Period: First Wear Period (8 -0/+3 Days)
Arm/Group | P1fA, Then AMfA | AMfA, Then P1fA
Started | 56; 112 eyes | 58; 116 eyes
Completed | 55; 110 eyes | 58; 116 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Adverse Event | 1 | 0
Period: Second Wear Period (8 -0/+3 Days)
Arm/Group | P1fA, Then AMfA | AMfA, Then P1fA
Started | 55; 110 eyes | 58; 116 eyes
Completed | 54; 108 eyes | 58; 116 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | P1fA, Then AMfA | AMfA, Then P1fA | Total
Number analyzed (Participants) | 56 | 58 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (9.9) | 32.1 (10.3) | 32.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 39 | 70
  Male | 25 | 19 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 47 | 47 | 94
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 11 | 23
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 10 | 23
  White | 31 | 36 | 67
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 56 | 58 | 114

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Distance VA (logMAR) With Study Lenses
Description: Distance visual acuity (VA) was assessed with study lenses in place. VA was collected for each eye separately using logarithmic of the Minimum Angle of Resolution (logMAR) charts. A logMAR acuity of 0.0 corresponds to 20/20 Snellen acuity (normal visual acuity), with a negative value denoting better than 20/20 visual acuity.
Time Frame: Day 8 (-0/+3 days), each study lens type
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study with non-missing response
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- P1fA: Verofilcon A toric contact lenses worn bilaterally (in both eyes) during the first wear period or the second wear period, as randomized, for 8 -0/+3 days in a daily disposable modality
- AMfA: Etafilcon A toric contact lenses worn bilaterally (in both eyes) during the first wear period or the second wear period, as randomized, for 8 -0/+3 days in a daily disposable modality
Arm/Group | P1fA | AMfA
Number analyzed (Participants) | 112 | 110
Number analyzed (eyes) | 224 | 220
logMAR | -0.08 (0.006) | -0.07 (0.006)
Statistical Analysis 1: Comparison: P1fA vs AMfA; Test type: Non-Inferiority — Noninferiority in distance VA was declared if upper confidence limit was less than 0.05; Mixed effects repeated measures model; Within subject correlation due to eye and the crossover design were accounted for in the model; Least Squares Means Difference = -0.01, 95% CI 1-sided [upper limit -0.01], Standard Error of Mean 0.004 — Lens difference (P1fA minus AMfA)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 22 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- P1fA Ocular; P1fA Nonocular: Events reported in this group occurred while exposed to the verofilcon A toric contact lenses
- AMfA Ocular; AMfA Nonocular: Events reported in this group occurred while exposed to the etafilcon A toric contact lenses
Arm/Group | Pretreatment | P1fA Ocular | P1fA Nonocular | AMfA Ocular | AMfA Nonocular
All-Cause Mortality (participants affected / at risk) | 0/114 | 0/228 | 0/114 | 0/226 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/114 | 0/228 | 1/114 | 0/226 | 0/113
Other Adverse Events (participants affected / at risk) | 0/114 | 0/228 | 0/114 | 0/226 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pretreatment (N=114) | P1fA Ocular (N=228) | P1fA Nonocular (N=114) | AMfA Ocular (N=226) | AMfA Nonocular (N=113)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04908488/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT04908488/SAP_001.pdf